CLINICAL TRIAL: NCT05310344
Title: Albumin-bound Paclitaxel and Bevacizumab for Platinum-resistant Recurrent Epithelial Ovarian Cancer: A Single-arm, Multi-center, Phase II Clinical Study
Brief Title: Albumin-bound Paclitaxel and Bevacizumab for Platinum-resistant Recurrent Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALBPAC1
Record Dates: First submitted 2022-03-26; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Ovarian Carcinoma; Platinum-resistant Ovarian Cancer; Recurrent Ovarian Carcinoma; Albumin-bound Paclitaxel; Bevacizumab; Survival Outcomes; Adverse Events
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Albumin-Bound Paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with platinum-resistant recurrent epithelial ovarian cancer (Experimental)
  Interventions: Combination Product: Albumin-bound paclitaxel and bevacizumab

INTERVENTIONS:
Combination Product: Albumin-bound paclitaxel and bevacizumab — Patients will receive albumin-bound paclitaxel (260 mg/m2) and bevacizumab (7.5mg/kg) intravenously every 21 days. The total treatment periods are no more than 6 cycles.

SUMMARY:
This study is a prospective, multicenter, phase II clinical trial to evaluate the efficacy and safety of albumin-bound paclitaxel combined with bevacizumab for platinum-resistant recurrent epithelial ovarian cancer. Patients with platinum-resistant recurrent ovarian cancer who meet the inclusion criteria, and don't meet any of the exclusion criteria, are enrolled in the study. They will receive albumin-bound paclitaxel (260 mg/m2) and bevacizumab (7.5mg/kg) intravenously every 21 days. Treatment continue until disease progression, intolerable toxicity, or patient refusal. Objective response rates primary objective. Progression-free survival, overall survival, and safety are secondary objectives. The study will enroll a total of 50 patients.

ELIGIBILITY:
Inclusion Criteria

1. Aged 18~75 years old
2. Histologically confirmed platinum-resistant recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer
3. At least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2;
5. Sufficient bone marrow function;
6. Sufficient liver and renal function;
7. Patients of reproductive potential were required to take effective contraceptive measures for the duration of the study and had a negative serum or urine pregnancy test result; non-lactating women;
8. Patients had no disturbance of consciousness and volunteered to participate in the study.

Exclusion Criteria

1. Uncontrolled hypertension
2. Tumor invading vital blood vessels
3. With contraindications to chemotherapy
4. With uncontrolled infection
5. Patients had received anticancer therapy within 3 weeks before enrollment
6. Patients were allergic or intolerant to investigational drugs or its ingredients
7. Patients are not suitable for this trial as judged by investigators

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-27 (Actual); Primary Completion 2023-03-27 (Estimated); Study Completion 2024-03-27 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 24 months
  ORR is defined as the percentage of participants in the analysis population who have a complete or partial remission per RECIST 1.1

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 24 months
  PFS defined as the time the duration from date of enrollment to the first documented disease progression per RECIST v1.1, or death due to any cause, whichever occurs first
Overall survival | 36 months
  Overall survival is defined as the duration from date of enrollment to the date of death from any cause
Adverse Events | 36 months
  Adverse event (AE), Treatment emergent adverse event (TEAE), Serious adverse event (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China